CLINICAL TRIAL: NCT04377828
Title: Evaluation of the Improvement of Pigmented Skin Lesions in Patients With Mastocytosis After Performing 2 Sessions of Pigment Laser : Pilot Study Conducted at a Reference Centre Mastocytoses (LaserMasto)
Brief Title: Improvement of Pigmented Skin Lesions in Patients With Mastocytosis After Performing 2 Sessions of Pigment Laser
Acronym: LaserMasto
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/19/0515; 2020-A00421-38 (Other: ID-RCB)
Record Dates: First submitted 2020-04-28; First posted 2020-05-06 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Cutaneous Mastocytosis
Keywords: Cutaneous mastocytosis; laser
MeSH Terms: conditions — Mastocytosis, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser intervention (Experimental): 1 to 2 sessions of pigment laser1
  Interventions: Device: Pigment laser

INTERVENTIONS:
Device: Pigment laser — one to two session of pigment laser (532 nm)

SUMMARY:
Cutaneous mastocytosis can be isolated or associated with systemic involvement. Urticaria pigmentosa affects around 80 to 85% of adult patients with cutaneous mastocytosis. It is also frequently present in patients with mastocytosis associated with systemic involvement (80% of patients in our experience).

This skin damage is one of the causes of deterioration in quality of life in patients with mastocytosis, through the loss of self-esteem, due to the appearance of lesions. However there are not treatment for urticaria pigmentosa.

Skin involvement in mastocytosis is linked to the accumulation of abnormal mast cells in the dermis. However, the mast cells are not pigmented and the brown-brown color characteristic of Urticaria pigmentosa is explained by melanin pigmentation of the epidermal basal layer.

DETAILED DESCRIPTION:
Cutaneous mastocytosis can be isolated or associated with systemic involvement. Urticaria pigmentosa affects around 80 to 85% of adult patients with cutaneous mastocytosis. It is also very frequently present in patients with mastocytosis associated with systemic involvement (80% of patients in our experience).

This skin damage is one of the causes of deterioration in quality of life in patients with mastocytosis, through the loss of self-esteem, due to the appearance of lesions. However ,there is not a treatment for urticaria pigmentosa.

Skin involvement in mastocytosis is linked to the accumulation of abnormal mast cells in the dermis. However, the mast cells are not pigmented and the brown-brown color characteristic of pigmentary urticaria is explained by melanin pigmentation of the epidermal basal layer. This characteristic is often described on skin biopsies of pigmentary urticaria analyzed in hematoxilin-eosin.

The 532 nm Q-Switched laser is known to improve lesions characterized by the presence of melanin pigment in the basal layer of the epidermis, with very little risks. This later is explained by the reduced penetration of light at 532 nm into the skin and the emission time of the laser light which is very low (of the order of a few nanoseconds) for Q-Switched lasers. In the literature, 2 case reports report an efficiency of the laser at 532 nm in this indication in adults.

The hypothesis of this study is that 2 sessions of Q-switched laser could improve the skin lesions of urticaria pigmentosa, leading to an improvement in self-esteem.

ELIGIBILITY:
Inclusion Criteria:

* Patient with mastocytosis (diagnosis confirmed clinically according to international criteria)
* Patient with pigmented skin lesions, of moderate to very severe severity (by comparison with a 4-point photographic scale: light, moderate, severe and very severe)
* Major patient aged ≥ 18 years.
* Patient with social security coverage
* Patient having given written, free and informed consent to participate in the study

Exclusion Criteria:

* Patients with mastocytosis, without skin lesions
* Patient with pigmented skin lesions, only of mild severity (by comparison with a 4-point photographic scale: mild, moderate, severe and very severe)
* Patient with another cutaneous mastocytosis phenotype
* Patient treated by a treatment known as a cytoreductive for mastocytosis: alpha interferon, cladribine, imatinib, midostaurin or any cytoreductive treatment being evaluated by clinical trial in mastocytosis
* Patient under guardianship, or under curatorship, or not fluent in the French language or unable to understand and complete the study questionnaires
* pregnant or breastfeeding women
* Patients with tanned skin following photoexposure within 3 weeks of starting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Global clinical evolution of the skin M4 - Blind evaluator | Month 4
  Global clinical evolution with IGA " Improvement Global Assessment" (scale with 5 points : no improvement or aggravation/minimal improvement/moderate improvement/significant improvement/complete disappearance) by blind evaluator in month 4 versus baseline

SECONDARY OUTCOMES:
Global clinical evolution of the skin M1 - Blind evaluator | Month 1
  Global clinical evolution with IGA " Improvement Global Assessment" (scale with 5 points : no improvement or aggravation/minimal improvement/moderate improvement/significant improvement/complete disappearance) by blind evaluator in month 1 versus baseline
Global clinical evolution of the skin M9 - Blind evaluator | Month 9
  Global clinical evolution with IGA " Improvement Global Assessment" (scale with 5 points : no improvement or aggravation/minimal improvement/moderate improvement/significant improvement/complete disappearance) by blind evaluator in month 9 versus baseline
Global clinical evolution of the skin M4 - Principal investigator | Month 4
  Global clinical evolution with IGA " Improvement Global Assessment" (scale with 5 points : no improvement or aggravation/minimal improvement/moderate improvement/significant improvement/complete disappearance) by the principal investigator in month 4 versus baseline
Global clinical evolution of the skin M1 - Principal investigator | Month 1
  Global clinical evolution with IGA " Improvement Global Assessment" (scale with 5 points : no improvement or aggravation/minimal improvement/moderate improvement/significant improvement/complete disappearance) by the principal investigator in month 1 versus baseline
Global clinical evolution of the skin M9 - Principal investigator | Month 9
  Global clinical evolution with IGA " Improvement Global Assessment" (scale with 5 points : no improvement or aggravation/minimal improvement/moderate improvement/significant improvement/complete disappearance) by the principal investigator in month 9 versus baseline
Severity of a targeted pigment skin lesion - M1 | Month 1
  the surface area of the target pigment skin lesion (mm2) versus baseline
Severity of a targeted pigment skin lesion - M4 | Month 4
  the surface area of the target pigment skin lesion (mm2) versus baseline
Severity of a targeted pigment skin lesion - M9 | Month 9
  the surface area of the target pigment skin lesion (mm2) versus baseline
Psychological impact - baseline | Baseline
  qualitative analysis of the patient verbatim after an interview
Psychological impact - Month 4 | Month 4
  qualitative analysis of the patient verbatim after an interview
Psychological impact - Month 9 | Month 9
  qualitative analysis of the patient verbatim after an interview
Patient satisfaction - Month 1 | month 1
  Global clinical evolution with IGA " Improvement Global Assessment" (scale with 5 points : no improvement or aggravation/minimal improvement/moderate improvement/significant improvement/complete disappearance) by patient versus baseline
Patient satisfaction - Month 4 | month 4
  Global clinical evolution with IGA " Improvement Global Assessment" (scale with 5 points : no improvement or aggravation/minimal improvement/moderate improvement/significant improvement/complete disappearance) by patient versus baseline
Patient satisfaction - Month 9 | month 9
  Global clinical evolution with IGA " Improvement Global Assessment" (scale with 5 points : no improvement or aggravation/minimal improvement/moderate improvement/significant improvement/complete disappearance) by patient versus baseline
global patient satisfaction | month 9
  Analog visual scale from 0 to 10
Pigment laser tolerance | Day 1
  Analog visual scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Christina BULAI LIVIDEANU, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Larrey Hospital - Toulouse University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No